CLINICAL TRIAL: NCT07111299
Title: Clinical Evaluation of Hair Loss, Hair Growth, and Skin Improvement in Human Volunteers Following a Double-blind, Placebo-controlled, 1:1 Randomized Trial of 'Olistic Next Women'
Brief Title: Clinical Evaluation of a Nutraceutical Supplement for Hair Growth, Hair Loss and Skin Improvement in Human Volunteers Versus Placebo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olistic Research Labs S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-ON-03
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Early Female Pattern Hair Loss (FPHL)
MeSH Terms: interventions — Minerals; Plant Extracts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Product Arm (Active Comparator)
  Interventions: Dietary Supplement: Drinkable multifactorial food supplement containing vitamins, minerals, plant extracts, and other bioactive compounds, formulated to support hair growth and scalp health in women.
- Placebo Arm (Placebo Comparator)
  Interventions: Other: Placebo Control

INTERVENTIONS:
Dietary Supplement: Drinkable multifactorial food supplement containing vitamins, minerals, plant extracts, and other bioactive compounds, formulated to support hair growth and scalp health in women. — Drinkable multifactorial food supplement in liquid form, administered once daily in a 25 mL single-dose vial, for a duration of 180 days. The formulation contains a combination of vitamins, minerals, plant extracts, amino acids, and other bioactive compounds designed to support hair growth and scalp health in women.
  Arms: Active Product Arm
Other: Placebo Control — Drinkable formulation consisting of an excipient formulation designed to mimic the organoleptic properties of the active product, reproducing its color and texture while achieving a highly similar taste profile.
  Arms: Placebo Arm

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of Olistic Next Women, a nutraceutical supplement, in women experiencing beginning of FPHL.

This 6-month, double-blind, placebo-controlled, 1:1 randomized clinical trial investigates whether daily supplementation with Olistic Next Women leads to significant improvements in hair parameters compared to placebo. The study also monitors the tolerability and safety of the product throughout the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50-65.
* Volunteers with initial FPHL. (Images will be sent to a dermatologist for assessment).
* Commitment not to use systemic, topical, or oral products with an effect similar to that of the product to be evaluated throughout the study period.
* Do not change the daily routine regarding the use of cosmetic products and eating habits.
* Commitment to comply with all protocol requirements specified in the subject information sheet.
* Availability to comply with all study visits.

Exclusion Criteria:

* Allergy or reactivity to some of the components of the product, or a product with similar category than tested one.
* Women who have undergone dermatological treatment for hair loss (PRPs, mesotherapy, etc.) or hair transplant.
* Scalp diseases: cicatricial alopecia, alopecia areata, folliculitis decalvans, psoriasis, moderate severe seborrheic dermatitis, eczema, cancer, etc.
* Women who present alopecia because of a medical illness (hypothyroidism, anemia, lupus, etc.).
* Relevant cutaneous marks in the experimental areas, which could interfere with the measurements (scars, sunburns, etc.).
* In-use relevant pharmacological or hormonal treatment (eg. valproic acid, carbamazepine, phenytoin).
* Women with thyroid alteration (hyper- or hypothyroidism)
* Women who have previously participated in similar studies or who have used anti-hair loss products in the last 3 months.
* Women who are being treated with anticoagulants, antifungals, anxiolytics, amphetamines, retinoids, iron, antithyroid, anticonvulsants, beta blockers and/or ACE inhibitors, minoxidil, finasteride, etc.
* Women who started hormonal treatment (oral or topical contraceptives) in the 6 months prior to the start of the study.
* Women who started taking any drug chronically less than 6 months before the start of the study (they should have a stable situation with the medication over 6 months).
* Modification of the usual diet: low-calorie diet, Atkins diet, etc.
* Pregnant, postpartum (6 months) or breastfeeding women, or who intend to get pregnant during the duration of the study.
* Evidence of systemic diseases (e.g. cardiac disease, psychiatric disease, etc.) or gastrointestinal diseases.
* Serious conditions or illnesses that, in the opinion of the researcher, may be aggravated by participation in the study or that put the development of the study at risk.
* Planned hairstyle changes throughout the study
* Presence of skin diseases or melanomas.
* Forecast of change of routine or relevant way of life, during the period of study.
* Other exclusion criteria to be added by the customer.
* Women who have gone dermatological treatment, that they have introduced minoxidil (oral or topical) at least 6 months prior, and antiandrogens (e.g. finasteride) at least 12 months before the start of the study.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Increase in hair density | From enrollment to the end of treatment at 180 days.
  From phototrichogram on the Sagittal midline area of the scalp

SECONDARY OUTCOMES:
Change in hair shedding | From enrollment to the end of treatment at 180 days.
  Hair shedding will be assessed by collecting shed hairs during a standardized washing and combing procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Bionos Biotech Clínica, Valencia, Spain